CLINICAL TRIAL: NCT02769091
Title: A 24-Week, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of 80 mg TEV-45478 Once Daily as Treatment in Adult Patients With Nonalcoholic Steatohepatitis (NASH) Who Also Have Type 2 Diabetes Mellitus - GN
Brief Title: A Study in Adult Patients With Nonalcoholic Steatohepatitis Who Also Have Type 2 Diabetes
Acronym: NASH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV45478-IMM-20019
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Nonalcoholic Steatohepatitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEV-45478 (Experimental): 80 mg (2x40mg) tablets once daily for up to 24 weeks
  Interventions: Drug: TEV-45478
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-45478 — 80 mg (2x40mg) tablets once daily for up to 24 weeks
  Arms: TEV-45478
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of TEV-45478, as compared with placebo, on liver health and liver fat content in patients with T2DM who also have Nonalcoholic Steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* The patient is female or male and aged 18 to 65 years, inclusive with a history of Type 2 Diabetes Mellitus (T2DM) and on stable medication for diabetes or insulin or a combination thereof for at least 3 months prior to screening.
* The patient has a NASH Activity Score (NAS) of ≥4, with or without evidence of fibrosis, with a score of at least 1 in steatosis and lobular inflammation the subcomponents of NAS and a hepatocyte ballooning score of at least 1 score based on historical histological evaluation of liver biopsy within 12 months prior to randomization.
* The patient has a historical diagnosis of NASH, established no more than 12 months prior to randomization based on histology (liver biopsy).
* The patient has an ALT level at screening between 45 and 105 IU/L, inclusive, for women and between 55 and 120 IU/L, inclusive for men, at one other occasion during the 24-weeks prior to screening.
* The patient has an MRI determined liver fat fraction of equal to or higher than 6% at Screening

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The patient has a history of chronic liver disease other than NASH eg, chronic or acute hepatitis, autoimmune, viral (A, B, C), genetic hepatitis, drug induced hepatotoxicity, Wilson's disease, alcoholic liver diseases, or any other non-NASH active liver disease.
* The patient has active cancer or a history of a malignant disease (except basal cell carcinoma of the skin) within 5 years prior to screening or any history of bladder cancer.
* The patient had an unstable metabolic condition (ie, with a history of weight loss or weight gain of >5 kg within 24 weeks prior to screening)
* The patient has a history of bariatric surgery within 5 years prior to screening.
* The patient has received mercaptopurine or azathioprine previously within 1 year prior to screening
* The patient has taken within 7 days prior to the first dose of study drug (or is anticipated to take during the study) anticholinergic or other drugs known to affect gastrointestinal (GI) motility, proton-pump inhibitors, or other drugs known to affect gastric acidity or use of allopurinol.
* The patient has received oral antibiotics within the last 4 weeks prior to randomization (day 1).
* The patient has received treatment within the last 30 days with any drugs known to induce or inhibit endogenous hepatic drug metabolism (eg, barbiturates, phenothiazines, cimetidine, carbamazepine) or anti-coagulant therapy (eg, heparin, warfarin, acenocoumarol).
* The patient has Type 1 Diabetes Mellitus (T1DM) or poorly controlled T2DM
* The patient has a body mass index (BMI) <25 kg/m2.
* The patient has a history of diabetic gastroparesis or has had gastric bypass surgery within the last 5 years.
* The patient has a history of pancreatitis.
* The patient has a history of persistent intestinal obstruction, bowel perforation, uncontrolled GI bleed or abdominal abscess or infection or toxic megacolon or inflammatory bowel disease (IBD)
* The patient has a history of coronary angioplasty, coronary stent placement, coronary bypass surgery, unstable angina, myocardial infarction, transient ischemic events, or stroke within 24-weeks prior to screening.
* The patient is classified as Class II-IV via New York Heart Association
* The patient has a history of drug abuse (defined as illicit drug use) or a history of excessive alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day for women or 3 alcoholic drinks per day for men) within 1 year prior to the screening visit.

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
serum Alanine Transaminase (ALT) levels response, defined as ALT value within reference range of <35 IU/L for women and <40 IU/L for men | Week 24
liver fat response, defined as a reduction of ≥6% at week 24 compared to screening by the MRI-Proton Density Fat Fraction (PDFF) | Week 24
Percentage of Participants with Adverse Events | 24 weeks

SECONDARY OUTCOMES:
percent change from baseline in ALT | Baseline, Week 24
percent change from baseline in ALT | Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24 (or early withdrawal)
percent change from baseline in Aspartate Aminotransferase (AST) | Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24 (or early withdrawal)
change from baseline in AST | Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24 (or early withdrawal)
change from baseline in ALT | Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24 (or early withdrawal)
Change from baseline in glycosylated hemoglobin ((HbA1c) | Baseline, Weeks 4, 12, and 24 (or early withdrawal)
Change from baseline in liver fibrosis measured using transient elastography (with Fibroscan) | Baseline, Week 24 (or early withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.